CLINICAL TRIAL: NCT04502316
Title: Real-World Experience -- Barostim™ Advancing the Level of Clinical Evidence (REBALANCE Registry) A Post-Market Registry With the Barostim™ System
Brief Title: Real-World Experience - Barostim™ Advancing the Level of Clinical Evidence (REBALANCE Registry)
Status: Active, not recruiting | Type: Observational
Sponsor: CVRx, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 360059-001
Record Dates: First submitted 2020-07-30; First posted 2020-08-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Barostim™ System — Implantation of the Barostim™ System

SUMMARY:
The purpose of this registry is to develop valid scientific evidence of the safety and benefit of Barostim Therapy in the commercial setting in patients with heart failure with reduced ejection fraction (HFrEF) that were recently implanted with the Barostim System.

DETAILED DESCRIPTION:
Summary:

The CVRx REBALANCE Registry includes patients who have been implanted with the Barostim System. Up to 5,000 patients will be enrolled. Data should be obtained from evaluations taken prior to implant, at implant, and every six months after device implant, up to the 36-month visit at which time each patient will be exited from the registry.

Enrollment data are collected retrospectively after consent and Barostim implant; post-enrollment data are collected prospectively from standard of care follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients can be included in the registry if they were implanted with a de novo Barostim System. Patients must sign an informed consent form after implantation with the Barostim System in order to participate in the registry.

Indications:

The Barostim System is indicated for the improvement of symptoms of heart failure - quality of life, six-minute hall walk and functional status - for patients who remain symptomatic despite treatment with guideline-directed medical therapy, are NYHA Class III or Class II (who had a recent history of Class III), have a left ventricular ejection fraction ≤ 35%, a NT-proBNP < 1600 pg/ml and excluding patients indicated for Cardiac Resynchronization Therapy (CRT) according to AHA/ACC/ESC guidelines.

Contraindications:

* Bilateral carotid bifurcations located above the level of the mandible
* Baroreflex failure or autonomic neuropathy
* Uncontrolled, symptomatic cardiac bradyarrhythmias
* Carotid atherosclerosis that is determined by ultrasound or angiographic evaluation greater than 50%
* Ulcerative plaques in the carotid artery as determined by ultrasound or angiographic evaluation
* Known allergy to silicone or titanium

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients can be included in the registry if they were implanted with a de novo Barostim System.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-06-26 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this post-market registry is to develop valid scientific evidence of the safety and benefit of Barostim Therapy in the commercial setting in patients that were recently implanted with the Barostim System. | 36 months post-implant

CONTACTS AND LOCATIONS:
Locations (46):
- United States (46):
  - Grandview Medical Center, Birmingham, Alabama
  - Chan Heart Rhythm Institute, Mesa, Arizona
  - Akil Loli Consulting LLC, Phoenix, Arizona
  - Cabrillo Cardiology Research Group, Oxnard, California
  - COR Healthcare Medical Associates, Torrance, California
  - Aurora Denver Cardiology Associates, Aurora, Colorado
  - South Denver Cardiology Associates, P.C., Littleton, Colorado
  - Medstar Health Research Insitutute, Washington D.C., District of Columbia
  - The George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Orlando Cardiac & Vascular Specialists, Altamonte Springs, Florida
  - Orlando Heart and Vascular Institute, Altamonte Springs, Florida
  - Lakewood Cardiovascular, Bradenton, Florida
  - AMA Heart and Vascular, Bradenton, Florida
  - Cardiovascular Solutions Institute, Bradenton, Florida
  - Cardiac Care Group, Cape Coral, Florida
  - Daytona Heart Group, Daytona Beach, Florida
  - Florida Heart Rhythm Specialists, Fort Lauderdale, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Premier Cardiology & Vascular Associates, Maitland, Florida
  - University of Miami, Miami, Florida
  - Naples Heart Rhythm Specialists, PA, Naples, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Sarasota Memorial Research Institute (Sarasota Memorial Hospital), Sarasota, Florida
  - University of South Florida, Tampa, Florida
  - Howard T. Tee, M.D., F.A.C.C., F.A.C.P., Vero Beach, Florida
  - Florida Cardiology (Guardian Research Organization, LLC), Winter Park, Florida
  - University of Chicago, Chicago, Illinois
  - Cardiovascular Medicine, Moline, Illinois
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Capitol Cardiology Associates, Lanham, Maryland
  - HeartPlus Diagnostic Center, Jackson, Mississippi
  - DeGregorio Cardiology, Glen Ridge, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Cardio Vascular Health Associates, South River, New Jersey
  - Capital Cardiology, Albany, New York
  - Marian David, M.D., P.C, Kew Gardens, New York
  - Adam Budzikowski PC, Maspeth, New York
  - Advanced Cardiac Care, Ozone Park, New York
  - Cone Health, Greensboro, North Carolina
  - Stern Cardiovascular, Germantown, Tennessee
  - Austin Heart, Austin, Texas
  - Baylor Scott & White Research Institute, Dallas, Texas
  - Centra Heart & Vascular Institute, Lynchburg, Virginia
  - Carient Heart & Vascular, Manassas, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin

IPD SHARING:
Plan to Share IPD: No